CLINICAL TRIAL: NCT02212834
Title: Comparative Effectiveness of Surveillance Modalities in Breast Cancer Survivors
Brief Title: Surveillance Imaging Modalities for Breast Cancer Assessment
Acronym: SIMBA
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Dartmouth College (Other); Harvard Pilgrim Health Care (Other); University of North Carolina, Chapel Hill (Other); University of California, San Francisco (Other); University of Wisconsin, Madison (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CE-1304-6656
Record Dates: First submitted 2014-03-21; First posted 2014-08-08 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Surveillance; Imaging; Comparative; Effectiveness
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mammograms: Surveillance mammograms in women with a personal history of breast cancer
- Breast MRI: Surveillance breast Magnetic Resonance Imaging (MRI) in women with a personal history of breast cancer

SUMMARY:
The purpose of this study is to determine the effectiveness of surveillance breast MRI compared to mammography alone in women with a personal history of breast cancer

DETAILED DESCRIPTION:
Our overall aim is to find out how well MRI works compared with mammography for surveillance in women who have previously had breast cancer. Specifically, our goals are to:

1. Understand doctors' and patients' experiences with surveillance mammography and MRI
2. Provide evidence on which outcomes are more or less likely to occur
3. Develop patient decision aids to help women and their doctors choose the surveillance method that is right for them

How we will conduct the study: We will work with patients, doctors, policy makers, advocacy groups, and researchers to improve surveillance for women who have a personal history of breast cancer. Through focus groups with patients and interviews with doctors, we will gain insights into women's experience with surveillance mammography and MRI. We will also compare mammography to MRI using data from the Breast Cancer Surveillance Consortium-the largest collection of breast cancer surveillance data in the nation. We will use data from more than 13,000 women diagnosed with breast cancer between 2005 and 2012 to determine how well each test works. We will measure the tests' effectiveness at finding second cancers, and estimate the likelihood of different outcomes. We will also determine whether one test appears to work better than the other to detect second breast cancers among different groups of women. We will then develop patient decision aids to help women and their doctors make more-informed choices about surveillance.

What we hope to achieve: We hope this study will improve medical decision making and care for the 3 million women in the United States who have a history of breast cancer. Specifically, our results will help women and their doctors make clearer, better choices about the surveillance method that is right for them.

ELIGIBILITY:
Inclusion Criteria: Surveillance imaging exams in women included in the Breast Cancer Surveillance Consortium who are 18+ years of age at the the of a Stage 0-III incident breast cancer diagnosis between January 1, 2005 and December 31, 2012.

-

Exclusion Criteria:

* Women with a diagnosis of lobular carcinoma in situ
* Women with missing cancer staging data from Surveillance, Epidemiology and End Results (SEER) Program records
* Women with Stage 4 breast cancer at time of diagnosis
* Women with a diagnosis of a second breast cancer event within six months of the primary diagnosis
* Women who die within six months of primary diagnosis
* Women who have had a double mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surveillance imaging exams in women included in the Breast Cancer Surveillance Consortium who are 18+ years of age at the the of a Stage 0-III incident breast cancer diagnosis between January 1, 2005 and December 31, 2012.
Sampling Method: Probability Sample
Enrollment: 36444 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Wernli, PhD, Principal Investigator — Group Health Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson DS, Bush MT, Brandzel S, Wernli KJ. The patient voice in research-evolution of a role. Res Involv Engagem. 2016 Feb 22;2:6. doi: 10.1186/s40900-016-0020-4. eCollection 2016. PMID 29062507
- [Background] Henderson LM, Ichikawa L, Buist DSM, Lee JM, Bush M, Johnson D, Onega T, Nekhlyudov L, Kerlikowske K, Miglioretti DL, Sprague BL, Wernli KJ. Patterns of Breast Imaging Use Among Women with a Personal History of Breast Cancer. J Gen Intern Med. 2019 Oct;34(10):2098-2106. doi: 10.1007/s11606-019-05181-6. Epub 2019 Aug 13. PMID 31410813
- [Result] Wernli KJ, Ichikawa L, Kerlikowske K, Buist DSM, Brandzel SD, Bush M, Johnson D, Henderson LM, Nekhlyudov L, Onega T, Sprague BL, Lee JM, Lehman CD, Miglioretti DL. Surveillance Breast MRI and Mammography: Comparison in Women with a Personal History of Breast Cancer. Radiology. 2019 Aug;292(2):311-318. doi: 10.1148/radiol.2019182475. Epub 2019 Jun 4. PMID 31161975
- See also: SIMBA Decision tool — https://www.artefactgroup.com/work/simba-breast-cancer-decisions-aid/
- See also: Video of impact of patient engagement in research — https://vimeo.com/154765251
- See also: Home page for the Breast Cancer Surveillance Consortium — https://www.bcsc-research.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort analysis of women with one or more observed breast cancer surveillance exams and primary cancer diagnosis between 2003 and 2012
Pre-assignment Details: Not a clinical trial. Analyses were conducted with the entire population who met study criteria. Unit of analysis was surveillance exam.
Units Other Than Participants: exams
Groups:
- Breast MRI: Surveillance Magnetic Resonance Imaging (MRI) in women with a personal history of breast cancer
Period: Overall Study
Arm/Group | Mammograms | Breast MRI
Started | 33938; 33,938 exams | 2506; 2,506 exams
Completed | 33938; 33,938 exams | 2506; 2,506 exams
Not Completed | 0; NA exams | 0; NA exams

BASELINE CHARACTERISTICS:
Population: Characteristics at time of surveillance exam
Units Other Than Participants: surveillance exams
Groups:
- Total: Total of all reporting groups
Arm/Group | Mammograms | Breast MRI | Total
Number analyzed (Participants) | 33,938 | 2,506 | 36444
Number analyzed (surveillance exams) | 33938 | 2506 | 36444
Age, Customized [Count of Units; unit: surveillance exams]
  Age at exam: 18 - 39 years | 388 | 153 | 541
  Age at exam: 40 - 49 years | 3,635 | 574 | 4209
  Age at exam: 50 - 59 years | 8,626 | 1,005 | 9631
  Age at exam: 60 - 69 years | 9,852 | 632 | 10484
  Age at exam: 70 - 79 years | 7,167 | 133 | 7300
  Age at exam: > or = 80 years | 4,270 | 9 | 4279
Sex: Female, Male [Count of Units; unit: surveillance exams]
  Female | 33,938 | 2,506 | 36444
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Units; unit: surveillance exams]
  Race/ethnicity at time of exam: White, non-hispanic | 26,717 | 2,069 | 28786
  Race/ethnicity at time of exam: Black, non-hispanic | 2,862 | 62 | 2924
  Race/ethnicity at time of exam: Hispanic | 1,042 | 67 | 1109
  Race/ethnicity at time of exam: Asian or Pacific Islander | 2,583 | 219 | 2802
  Race/ethnicity at time of exam: Mixed or Other | 657 | 88 | 745
  Race/ethnicity at time of exam: Missing | 77 | 1 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Breast Cancers Detected
Description: Number of second breast cancers detected in the 12 months after surveillance mammogram or breast MRI
Time Frame: 12 months post surveillance exam
Measure: Number; unit: cancers detected
Units Other Than Participants: exams
Arm/Group | Mammograms | Breast MRI
Number analyzed (Participants) | 33,938 | 2,506
Number analyzed (exams) | 33938 | 2506
cancers detected | 279 | 27

ADVERSE EVENTS:
Description: This study was not a clinical trial. It was a cohort analysis, with no study intervention and no participant contact. Adverse events are not applicable.
Arm/Group | Mammograms | Breast MRI
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was not a clinical trial. It was a cohort analysis of existing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No